CLINICAL TRIAL: NCT02091154
Title: Evaluating the Impact on Lunch Sales and Consumption of New School Lunch Guidelines and Behavioral Interventions in NYC Schools
Brief Title: How Environmental Interventions Influence Behavior in School Lunchrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 1202002824
Record Dates: First submitted 2014-03-03; First posted 2014-03-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Child Behavior; Adolescent Behavior; Health Behavior
Keywords: Food Intake Regulation; Fruit; Vegetable
MeSH Terms: conditions — Child Behavior; Adolescent Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- USDA Regulations Only (Experimental): Implement USDA Regulations in assigned school cafeterias during the intervention period.
  Interventions: Behavioral: USDA Regulations
- USDA Regulations and Marketing Kit (Experimental): Implement new USDA regulations in assigned schools along with the Marketing Kit during the intervention period.
  Interventions: Behavioral: USDA Regulations; Behavioral: Marketing Kit
- USDA Regulations and SLM (Experimental): Implement USDA Regulations and Smarter Lunchrooms Makeover in assigned schools during intervention period.
  Interventions: Behavioral: USDA Regulations; Behavioral: Smarter Lunchrooms Makeover (SLM)
- Control (No Intervention): Schools assigned to this intervention made no changes to their lunchroom or menus.

INTERVENTIONS:
Behavioral: USDA Regulations — Implement new USDA regulations assigned school cafeterias.
  1. Fruit or vegetable on every tray
  2. Meet requirements for vegetable varieties
  3. 50% of all grains must be whole grain
  4. Milk must be 1% or skim; flavored milk must be skim
  Arms: USDA Regulations Only; USDA Regulations and Marketing Kit; USDA Regulations and SLM
Behavioral: Marketing Kit — This marketing tool kit is designed to encourage purchasing of school lunches. The marketing tool kit included the following components:
  1. 56''x72'' vinyl sign with the words "[school mascot] Cafe"
  2. 8.5''x11'' signs describing the foods offered on a specific day
  3. 2''x4'' signs used to name all foods. These were to be placed in a visible location near the corresponding food.
  4. Magnetic board displaying a tray onto which magnets shaped as food can be placed to show what foods were being offered during a specific lunch shift.
  Arms: USDA Regulations and Marketing Kit
Behavioral: Smarter Lunchrooms Makeover (SLM) — Implement three basic Smarter Lunchrooms techniques. It consists of the following components:
  1. Place fruit in an attractive bowl or serving dish and set on two places on the line. One of the places should be at or near the register.
  2. Give all vegetables descriptive names and write or type them on a 2''x4'' card. These cards should be visible and placed near the corresponding food.
  3. Make white milk the most prominent milk in the milk coolers by making it the most available milk and easiest to take.
  Arms: USDA Regulations and SLM

SUMMARY:
The investigators hypothesize that the new United States Department of Agriculture (USDA) regulations for lunches served as part of the National School Lunch Program will decrease the percentage of enrolled students purchasing lunch, increase the percentage of children taking fruit and vegetables, decrease the percentage of fruit and vegetable servings being thrown away, and increase the total number of fruit and vegetable servings eaten.

The investigators also hypothesize that when the regulations are in force, simple behavioral interventions can counteract the potentially negative impact on lunch sales and consumption. In other words, implementing the regulations and behavioral interventions together, the percentage of enrolled students taking a school lunch will increase at least back to baseline levels, the percentage of children taking fruits and vegetables will increase, the percentage of fruit and vegetable servings wasted will decrease, and the total number of fruit and vegetable servings eaten will increase.

DETAILED DESCRIPTION:
This study was conducted in 43 schools in the New York City (NYC) School district in the spring of 2012. The new regulations for school lunches were scheduled to roll out nationally in the fall of the same year, so this study was designed to provide an indication of the impact the new regulations would have.

In addition to the regulations, the investigators also tested additional behavioral interventions, in conjunction with the regulations, to determine how the behavioral interventions might offset, or magnify, the impacts of the regulations.

ELIGIBILITY:
Inclusion Criteria:

* Public schools with any combination of grades K-12

Exclusion Criteria:

* No point of sale system in school
* Satellite school
* Feeder school

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in percent fruit or vegetable waste by student | Six months
  In the twelve schools, tray waste data were collected twice in April 2012 and once in May 2012. Results were generated and reported in September 2012.

SECONDARY OUTCOMES:
Change in lunch sales | Six months
  Lunch sales data were collected each school day in the 43 schools from March through May 2012. Results were generated and reported in September 2012.

OTHER OUTCOMES:
Change in servings of fruits and vegetables taken | Six months
  Each school cafeteria keeps records on the number of servings of each food served during a lunch period. These data were collected each day in the 43 schools from March through May 2012. Results were generated and reported in September 2012.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Brumberg, BA, Principal Investigator — Cornell University; Kathryn Hoy, RD, MFN, Principal Investigator — Cornell University; David Just, PhD, Study Chair — Cornell University; Brian Wansink, PhD, Study Director — Cornell University; Andrew Hanks, PhD, Principal Investigator — Cornell University
Locations (1):
- New York City School District, New York, New York, United States

REFERENCES:
- [Background] Hanks AS, Wansink B, Just DR. Reliability and accuracy of real-time visualization techniques for measuring school cafeteria tray waste: validating the quarter-waste method. J Acad Nutr Diet. 2014 Mar;114(3):470-474. doi: 10.1016/j.jand.2013.08.013. Epub 2013 Oct 14. PMID 24135053
- [Background] Hanks AS, Just DR, Wansink B. Smarter lunchrooms can address new school lunchroom guidelines and childhood obesity. J Pediatr. 2013 Apr;162(4):867-9. doi: 10.1016/j.jpeds.2012.12.031. Epub 2013 Feb 22. PMID 23434267
- [Background] Wansink B, Just DR, Hanks AS, Smith LE. Pre-sliced fruit in school cafeterias: children's selection and intake. Am J Prev Med. 2013 May;44(5):477-80. doi: 10.1016/j.amepre.2013.02.003. PMID 23597811
- [Background] Hanks AS, Just DR, Smith LE, Wansink B. Healthy convenience: nudging students toward healthier choices in the lunchroom. J Public Health (Oxf). 2012 Aug;34(3):370-6. doi: 10.1093/pubmed/fds003. Epub 2012 Jan 31. PMID 22294661